CLINICAL TRIAL: NCT02347163
Title: A Multicenter, Single-arm, Phase II Study to Evaluate the Activity of Pre-operative Zoledronate in Triple Negative Breast Cancer Patients, According to p53 Level
Brief Title: Pre-operative Zoledronate in Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study stopped prematurely due to the low accrual rate
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRFMN-BRC-6591
Record Dates: First submitted 2015-01-15; First posted 2015-01-27 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer
Keywords: triple neg; breast cancer; zoledronate; mevalonate pathway
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zoledronate (Experimental): Patients fulfilling the eligibility criteria will receive a pre-operative, single administration of zoledronate (4mg i.v.), 7 days before definitive breast surgery
  Interventions: Drug: Zoledronate

INTERVENTIONS:
Drug: Zoledronate — Patients fulfilling the eligibility criteria will be registered using a centralized system and will receive a pre-operative, single administration of zol (4mg i.v.), 7 days before definitive breast surgery .
  Other Names: Zometa

SUMMARY:
Recent evidences suggest that zoledronate (zol), one of the most used bisphosphonates (BPs) in the clinical setting for the prevention and treatment of bone metastasis in cancer patients, may have antitumor activity in early breast cancer in terms of improved disease free survival, overall survival and better response in BPs treated patients. BPs are mevalonate pathway inhibitors and one of the most intriguing hypothesis supporting their anticancer activity relies on the modulation of the mevalonate downstream metabolism. Biologically active mevalonate metabolites are involved in tumour cell proliferation and invasion and selected cancer subtypes may present a more pronounced mevalonate activity, able of maintaining an aggressive phenotype. The mevalonate pathway has deep impact on the function of YAP/TAZ, transcriptional regulators of tumour growth, and preclinical evidences suggest that BPs are able to interfere with YAP/TAZ expression, via mevalonate pathway. This study addresses the clinical role of BPs in triple negative breast cancer (TNBC) patients selected by the level of mevalonate pathway regulation, namely the p53 expression. This study is a multicenter single-arm, phase II study primarily aimed at assessing the anti-tumor activity of pre-operative zol measured through its effect on the Ki67 proliferative biomarker, in TNBC patients classified according to the p53 expression (high vs low p53 expression). Patients with newly diagnosed, untreated, operable TNBC, intended to definitive breast surgery and suitable for pre-operative therapy with zoledronate will receive a pre-operative, single administration of zol (4mg i.v.), 7 days before definitive breast surgery. Ki67 levels will be assessed in tumor samples collected at the time of diagnosis and after zoledronate treatment at the time of definitive surgery. The secondary objective of the study is to investigate the effect of zoledronate on critical genes/proteins related to p53 and mevalonate pathways, p53/PIN1 and YAP/TAZ, analyzed in the tumor tissue collected at the time of diagnosis and at definitive surgery. Zol safety profile will be evaluated by the NCI-CTCAE scale, version 4.0, and by the occurrence of serious adverse reactions. The total number of patients required is forty. The overall duration of the project is 32 months (30 months for accrual, followed by 2 months of follow-up after the recruitment of the last patient).

DETAILED DESCRIPTION:
Recent evidences suggest that zoledronate, one of the most used bisphosphonates (BPs) in the clinical setting for the prevention and treatment of bone metastasis in cancer patients, may have antitumor activity in early breast cancer. Notwithstanding some conflicting data, the majority of the clinical trials have shown some positive effects of BPs on patients outcome, reporting improved Disease Free Survival (DFS) and Overall Survival in mostly chemotherapy-naive premenopausal patients after a 3-year treatment with zoledronate and better DFS for immediate use of zoledronate in postmenopausal patients receiving adjuvant aromatase inhibitor treatment. Moreover, early breast cancer patients treated with neoadjuvant chemotherapy in combination with zoledronic acid showed better response compared with chemotherapy alone.

Even though different explanations have been proposed over-time, the exact mechanism of action of the anti-tumor activity of BPs is still not well understood. Basically, BPs are mevalonate pathway inhibitors and one of the most intriguing hypothesis supporting their anticancer activity relies on the modulation of the mevalonate downstream metabolism. Biologically active mevalonate metabolites are involved in tumour cell proliferation, survival, invasion and metastasis. Moreover, there is evidence that selected cancer subtypes may present a more pronounced mevalonate activity, able of maintaining an aggressive phenotype. Indeed, the mevalonate pathway has deep impact on the function of YAP/TAZ, transcriptional regulators of tumour growth. Preclinical evidences, suggest that BPs are able to interfere with YAP/TAZ expression, via mevalonate pathway. This study addresses the clinical role of BPs in triple negative breast cancer (TNBC) patients selected by the level of mevalonate pathway regulation, namely the p53 expression.

This study is a multicenter single-arm, phase II study primarily aimed at assessing the anti-tumor activity of pre-operative zoledronate measured through its effect on the Ki67 proliferative surrogate biomarker, in patients with TNBC classified according to the p53 expression (high vs low p53 expression). An high level of p53 is defined by IHC expression ≥30%, while a low level is defined by IHC expression <30%, as previously described. Patients with newly diagnosed, untreated, operable TNBC, intended to definitive breast surgery and suitable for pre-operative therapy will be registered using a centralized system and will receive a pre-operative, single administration of zoledronate (4mg i.v.), 7 days before definitive breast surgery . Ki67 levels will be assessed in core biopsy tumor samples collected at the time of diagnosis and after zoledronate treatment at the time of definitive surgery. Primary endpoint of the study is the proportion of responder patients, defined as those with at least 30% reduction in Ki67 at surgery with respect to core-biopsy analysis. The secondary objective of the study is to investigate the effect of zoledronate on critical genes/proteins related to p53 and mevalonate pathways, p53/PIN1 and YAP/TAZ, analyzed in the tumor tissue at the time of diagnosis (core biopsy) and at definitive surgery. The safety profile of zoledronate will be evaluated by the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) scale, version 4.0 and by the occurrence of serious adverse reactions. The total number of patients required is forty. The overall duration of the project is expected to be 32 months, divided as follows: 30 months for accrual, followed by 2 months of follow-up after the recruitment of the last patient, aimed to collect data on zoledronate safety and tolerability. The primary analysis will be conducted on the PP population which will include all patients registered, who received the dose of study treatment and underwent definitive breast surgery, with no major violations of the eligibility criteria or during study conduction. Proportion of responder patients, defined as those with at least 30% reduction in Ki67 at surgery with respect to core-biopsy analysis, will be presented as point estimate and 95% confidence intervals (95% CIs) for each group. Logistic regression techniques will be used to compare groups in univariate and multivariate model adjusted for ECOG-PS, sex and pre- and postmenopausal status. The results of this project may eventually contribute to unveil novel anticancer mechanism of action of BPs and new therapeutic options for triple negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-metastatic operable primary invasive TN breast cancer subjected to diagnostic core biopsy
* TNBC defined as HER2/ER/PgR negative receptors
* Ki67 and p53 expression determined by IHC
* Tumour tissue availability at time of diagnosis for IHC evaluation of p53/PIN1, YAP/TAZ and Ki67 protein expression and for RT-PCR molecular testing of critical genes: p53/PIN1, YAP/TAZ
* Age ≥ 18 years old
* ECOG (Eastern Cooperative Oncology Group) performance status ≤ 1
* Patients with reproductive potential. Female patients must have a negative serum pregnancy test within 7 days prior to start of trial. Patients must agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months (female patients) and 6 months (male patients) after discontinuation of treatment
* Written informed consent signed prior to enrolment according to ICH/GCP.

Exclusion Criteria:

* Presence of metastatic disease
* Clinical indication of debulking neo-adjuvant treatment
* Previous investigational treatment for any condition within 4 weeks from study registration
* Treatment with bisphosphonates, denosumab or other drug that, in the Investigator's judgment, affects bone metabolism
* Treatment with statins or other drugs that, in the Investigator's judgment, potentially affect the mevalonate pathway
* Any previous treatment for the currently diagnosed breast cancer, including radiation therapy, chemotherapy, biotherapy and/or hormonal therapy
* Inadequate bone marrow, hepatic or renal function including the following

  1. Hb< 9.0 g/dL, absolute neutrophil count < 1.5 x 109/L, platelets <100 x 109/L
  2. Total bilirubin > 1.5 x ULN, excluding cases where elevated bilirubin can be attributed to Gilberts Syndrome
  3. AST (SGOT), ALT (SGPT) > 2.5 x ULN Creatinine > 1.2 x ULN, calcium <8.6mg/dL
* Co-existing active infection or serious concurrent illness that, at the judgment of the investigator, contra-indicate the inclusion of the patient in the study
* Co-existing dental diseases that form a contraindication to the use of zol or need for immediate dental work
* Any medical or other condition that in the investigator's opinion renders the patient unsuitable for this study due to unacceptable risk
* Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary study assessment and procedures
* Anticipation of need for major surgical procedure during the course of the trial
* Known hypersensitivity to any excipients of zoledronate
* Pregnant or breast feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Assessment of zoledronate effect on Ki67 proliferative surrogate biomarker expression, according to p53 expression | 18 months
  The study is primarily aimed at assessing the anti-tumor activity of pre-operative zoledronate, measured through its effect on the Ki67 proliferative surrogate biomarker, in patients with TNBC selected according to the p53 expression (high vs low p53 expression). Primary endpoint of the study is the proportion of responder patients, defined as those with at least 30% reduction in Ki67 at surgery with respect to core-biopsy analysis. Prior to enrolment, the FFPE diagnostic core biopsy specimens will be analyzed by the study pathologist to determine the presence of invasive TNBC and the Ki67/p53 values. The Ki67/p53 evaluation will be then repeated after treatment at the time of definitive surgery

SECONDARY OUTCOMES:
Effect of zoledronate on critical genes/proteins related to p53 and mevalonate pathways, p53/PIN1 and YAP/TAZ (FFPE core biopsy will be tested for critical genes/proteins expression (by RT-PCR and IHC), including p53/PIN1 and YAP/TAZ) | 18 months
  The secondary endpoint of the study is aimed to investigate the effect of zoledronate on critical genes/proteins related to p53 and mevalonate pathways, p53/PIN1 and YAP/TAZ, analyzed at the time of diagnosis (core biopsy) and at definitive surgery (breast cancer resection). After enrolment, the FFPE core biopsy will be tested for critical genes/proteins expression (by RT-PCR and IHC), including p53/PIN1 and YAP/TAZ. The same evaluations will be performed after treatment, at the time of definitive surgery
Assessment of zoledronate safety (valuated by the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) scale, version 4.0 and by the occurrence of serious adverse reactions) | participants will be followed for AE occurrence from the informed consent signature to 2 months after study drug administration
  The safety profile of zoledronate will be evaluated by the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) scale, version 4.0 and by the occurrence of serious adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Zambelli, MD, Principal Investigator — Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
Locations (4):
- Italy (4):
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia, BS
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Oncologia 2 Istituto Oncologico Veneto IRCCS, Padua
  - Fondazione Salvatore Maugeri - IRCCS, Pavia

IPD SHARING:
Plan to Share IPD: No
The final clinical study report will be sent to the participating researchers

REFERENCES:
- [Background] Reis-Filho JS, Tutt AN. Triple negative tumours: a critical review. Histopathology. 2008 Jan;52(1):108-18. doi: 10.1111/j.1365-2559.2007.02889.x. PMID 18171422
- [Background] Lehmann BD, Bauer JA, Chen X, Sanders ME, Chakravarthy AB, Shyr Y, Pietenpol JA. Identification of human triple-negative breast cancer subtypes and preclinical models for selection of targeted therapies. J Clin Invest. 2011 Jul;121(7):2750-67. doi: 10.1172/JCI45014. PMID 21633166
- [Background] Gnant M, Mlineritsch B, Luschin-Ebengreuth G, Kainberger F, Kassmann H, Piswanger-Solkner JC, Seifert M, Ploner F, Menzel C, Dubsky P, Fitzal F, Bjelic-Radisic V, Steger G, Greil R, Marth C, Kubista E, Samonigg H, Wohlmuth P, Mittlbock M, Jakesz R; Austrian Breast and Colorectal Cancer Study Group (ABCSG). Adjuvant endocrine therapy plus zoledronic acid in premenopausal women with early-stage breast cancer: 5-year follow-up of the ABCSG-12 bone-mineral density substudy. Lancet Oncol. 2008 Sep;9(9):840-9. doi: 10.1016/S1470-2045(08)70204-3. Epub 2008 Aug 19. PMID 18718815
- [Background] Bundred NJ, Campbell ID, Davidson N, DeBoer RH, Eidtmann H, Monnier A, Neven P, von Minckwitz G, Miller JC, Schenk NL, Coleman RE. Effective inhibition of aromatase inhibitor-associated bone loss by zoledronic acid in postmenopausal women with early breast cancer receiving adjuvant letrozole: ZO-FAST Study results. Cancer. 2008 Mar 1;112(5):1001-10. doi: 10.1002/cncr.23259. PMID 18205185
- [Background] Coleman RE, Winter MC, Cameron D, Bell R, Dodwell D, Keane MM, Gil M, Ritchie D, Passos-Coelho JL, Wheatley D, Burkinshaw R, Marshall SJ, Thorpe H; AZURE (BIG01/04) Investigators. The effects of adding zoledronic acid to neoadjuvant chemotherapy on tumour response: exploratory evidence for direct anti-tumour activity in breast cancer. Br J Cancer. 2010 Mar 30;102(7):1099-105. doi: 10.1038/sj.bjc.6605604. Epub 2010 Mar 16. PMID 20234364
- [Background] Paterson AH, Anderson SJ, Lembersky BC, Fehrenbacher L, Falkson CI, King KM, Weir LM, Brufsky AM, Dakhil S, Lad T, Baez-Diaz L, Gralow JR, Robidoux A, Perez EA, Zheng P, Geyer CE Jr, Swain SM, Costantino JP, Mamounas EP, Wolmark N. Oral clodronate for adjuvant treatment of operable breast cancer (National Surgical Adjuvant Breast and Bowel Project protocol B-34): a multicentre, placebo-controlled, randomised trial. Lancet Oncol. 2012 Jul;13(7):734-42. doi: 10.1016/S1470-2045(12)70226-7. Epub 2012 Jun 14. PMID 22704583
- [Background] Ben-Aharon I, Vidal L, Rizel S, Yerushalmi R, Shpilberg O, Sulkes A, Stemmer SM. Bisphosphonates in the adjuvant setting of breast cancer therapy--effect on survival: a systematic review and meta-analysis. PLoS One. 2013 Aug 26;8(8):e70044. doi: 10.1371/journal.pone.0070044. eCollection 2013. PMID 23990894
- [Background] Holen I, Coleman RE. Anti-tumour activity of bisphosphonates in preclinical models of breast cancer. Breast Cancer Res. 2010;12(6):214. doi: 10.1186/bcr2769. Epub 2010 Dec 16. PMID 21176176
- [Background] Goldstein JL, Brown MS. Regulation of the mevalonate pathway. Nature. 1990 Feb 1;343(6257):425-30. doi: 10.1038/343425a0. PMID 1967820
- [Background] Freed-Pastor WA, Mizuno H, Zhao X, Langerod A, Moon SH, Rodriguez-Barrueco R, Barsotti A, Chicas A, Li W, Polotskaia A, Bissell MJ, Osborne TF, Tian B, Lowe SW, Silva JM, Borresen-Dale AL, Levine AJ, Bargonetti J, Prives C. Mutant p53 disrupts mammary tissue architecture via the mevalonate pathway. Cell. 2012 Jan 20;148(1-2):244-58. doi: 10.1016/j.cell.2011.12.017. PMID 22265415
- [Background] Wang Z, Wu Y, Wang H, Zhang Y, Mei L, Fang X, Zhang X, Zhang F, Chen H, Liu Y, Jiang Y, Sun S, Zheng Y, Li N, Huang L. Interplay of mevalonate and Hippo pathways regulates RHAMM transcription via YAP to modulate breast cancer cell motility. Proc Natl Acad Sci U S A. 2014 Jan 7;111(1):E89-98. doi: 10.1073/pnas.1319190110. Epub 2013 Dec 23. PMID 24367099
- [Background] Sorrentino G, Ruggeri N, Specchia V, Cordenonsi M, Mano M, Dupont S, Manfrin A, Ingallina E, Sommaggio R, Piazza S, Rosato A, Piccolo S, Del Sal G. Metabolic control of YAP and TAZ by the mevalonate pathway. Nat Cell Biol. 2014 Apr;16(4):357-66. doi: 10.1038/ncb2936. Epub 2014 Mar 23. PMID 24658687
- [Background] Piccolo S. LIF-ting Hippo averts metastasis. Nat Med. 2012 Oct;18(10):1463-5. doi: 10.1038/nm.2955. No abstract available. PMID 23042347
- [Background] Havrilesky L, Darcy kM, Hamdan H, Priore RL, Leon J, Bell J, Berchuck A; Gynecologic Oncology Group Study. Prognostic significance of p53 mutation and p53 overexpression in advanced epithelial ovarian cancer: a Gynecologic Oncology Group Study. J Clin Oncol. 2003 Oct 15;21(20):3814-25. doi: 10.1200/JCO.2003.11.052. PMID 14551300
- [Background] Wiltschke C, Kindas-Muegge I, Steininger A, Reiner A, Reiner G, Preis PN. Coexpression of HER-2/neu and p53 is associated with a shorter disease-free survival in node-positive breast cancer patients. J Cancer Res Clin Oncol. 1994;120(12):737-42. doi: 10.1007/BF01194273. PMID 7798300
- [Background] Dowsett M, Nielsen TO, A'Hern R, Bartlett J, Coombes RC, Cuzick J, Ellis M, Henry NL, Hugh JC, Lively T, McShane L, Paik S, Penault-Llorca F, Prudkin L, Regan M, Salter J, Sotiriou C, Smith IE, Viale G, Zujewski JA, Hayes DF; International Ki-67 in Breast Cancer Working Group. Assessment of Ki67 in breast cancer: recommendations from the International Ki67 in Breast Cancer working group. J Natl Cancer Inst. 2011 Nov 16;103(22):1656-64. doi: 10.1093/jnci/djr393. Epub 2011 Sep 29. PMID 21960707